CLINICAL TRIAL: NCT06528379
Title: Physical Activity Component of the Greek Interventional Geriatric Study to Prevent Cognitive Impairment and Disability (GINGER): Study Protocol and Feasibility of the Assessment
Brief Title: Physical Activity Component of the Greek Interventional Geriatric Study to Prevent Cognitive Impairment and Disability (GINGER)
Acronym: GINGER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Patras (Other)
Collaborators: University Hospital of Patras (Other); University Hospital of Crete (Other)
Responsible Party: Principal Investigator, Evdokia Billis, Professor in Physiotherapy, University of Patras
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GINGER_Physical Activity
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: People With Subjective Cognitive Impairement (SCI)
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical Activity intervention (Experimental): This Physical Activity intervention arm is a 6-month excercise protocol for SCI people, delivered 3 times per week, comprising of 2 supervised group-based exercise sessions & one home-based (unsupervised) one.
  The exercise programme is a progressive evidence-based tailored exercise regime comprising aerobic, resistance and balance exercises, applied at a moderate intensity (60-80% of targeted heart rate).
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity — The exercise programme is a 6-month progressive tailored-based exercise regime comprising
  * aerobic exercises (40-60%)
  * resistance exercises (20-40%)
  * balance with resistance exercises (20%) .
  This is peformed 3 times weekly, it is tailored to each individual but delivered in a small group-based manner. Two sessions are supervised by physiotherapist /exercise scientist and one session is unsupervised, home-based.

SUMMARY:
The Greek Interventional Geriatric Study to Prevent Cognitive Impairment and Disability (GINGER) is a six-month multimodal, multicenter study aimed at people with Subjective Cognitive Impairement (SCI).

One of the GINGER's interventional components is the Physcial Activity (PA) component, coordinated by the University of Patras.

This PA component's scope is to determine whether an enhanced individualized physical exercise intervention programme can improve cognitive changes, physical function, quality of life and wellbeing in people with subjective cognitive decline.

ELIGIBILITY:
Inclusion Criteria include people with:

* Subjective Cognitive Decline confirmed from the Subjctive Cognitive Decline Questionnaire (SCD - Q score >7)
* Absence of objective cognitive imparement as confirmed from cognitive assessment tests (i.e. MoCA, Trail A & B, Stroop, RCFT, FAS. )

Exclusion Criteri include people with:

* Mild Cognitive Impairement (MCI) or dementia
* Chronic psychiatric or neurological disorders affecting cognition (i.e. bipolar disorder, schizophrenia, MS, TBI, Parkinson's disease etc.)
* Unstable pathological diseases (i.e. uncontrolled hypothyrodism, athythmias, uncontrolled hypertension, high blood pressure at rest etc.)
* Recent (<6 month) surgery, which restrics active participation in exercise/physical activity
* inadequate knowledge of Greek

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Balance | Baseline, midway (12-weeks), post-intervention (6months) & follow-up (3 months)
  The Greek version of the Mini-BESTest (Mini-Balance Evaluation Systems Test) is used to assess the balance of each participant comprising four primary assessment balance categories (anticipatory, reactive postural control, sensory orientation, dynamic gait). The Mini-BESTest focuses primarily on dynamic balance and contains 14 different balancing tasks, each scored from 0 (lowest level of function) to 2 (highest level of function). Thus, overall scores range from 0 (lowest level of function) to 28 (highest level of function) and subsequent subscales are scored as: Anticipatory tasts (0-6), Reactive Postural Control (0-6), Sensory Orientation (0-6) & Dynamic Gait (0-10). Mini-BESTest takes about 10-15 minutes to be administered.
Upper limb muscle strength | Baseline, midway (12-weeks), post-intervention (6months) & follow-up (3 months)
  The Hand Grip Strength test is an objective, established and standardised measure of upper limb muscle strength, comprising a standard electronic hand dynamometer (Jamar) for measuring muscle strength of the hand (measured in kgs).
Lower limb muscle strength | Baseline, midway (12-weeks), post-intervention (6months) & follow-up (3 months)
  The lower limbs strength is measured using the 30 seconds Sit-to-Stand test, which is an objective, established and standardised measure of lower limb muscle strength. Participants are seated in the front part of a standard chair with their hands crossed in front of their chest, and they are asked to stand up completely (full extension of their knees) and sit back down to the chair as many times as possible during 30 seconds (measuring the repetitions).
Aerobic capacity | Baseline, midway (12-weeks), post-intervention (6months) & follow-up (3 months)
  The 2 Minute Walk Test is an established and objective test for measuring aerobic capacity. Participants are placed in a hallway of nine meters and are asked to cover as much ground as they can in two minutes (measured in meters).

SECONDARY OUTCOMES:
Fear of Falling | Baseline, midway (12-weeks), post-intervention (6months) & follow-up (3 months)
  The Greek version of the Falls Self-efficacy International Scale (FES-I_GREEK) is used to evaluate Fear of Falling. FES-I is a 16-item questionnaire with scores ranging from 16 to 64 points. Higher scores indicate higher fear and concern regarding falls.
Physical Function | Baseline, midway (12-weeks), post-intervention (6months) & follow-up (3 months)
  The International Physical Activity Questionnaire (IPAQ- 7) is used to evaluate physical function. IPAQ-7 is a 7-item questionnaire that calculates the physical activities taken place the last week (measured in METs).
Adherance to exercise | Baseline, midway (12-weeks), post-intervention (6months) & follow-up (3 months)
  The Exercise Adherance Rating Scale (EARS) is a validated and recently adapted into Greek outcome for measuring execise adhearance as well as the reasons of non-adhearing, comprising of 16 question items, exploring adhearance (6 question items) and reasons for adhearance/non-adhearance (10 items). Scores range from 0 (adherance) to 64 (non-adherance).

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - Laboratory of Clinical Physiotherapy and Research, Department of Physiotherapy, University of Patras, Pátrai, Achaia
  - Department of Psychiatry, School of Medicine, University of Patras, Pátrai

IPD SHARING:
Plan to Share IPD: Undecided
Yes, once we gather 50% of the data, we will be happy to share.